CLINICAL TRIAL: NCT02646657
Title: An Open Label Interventional Phase 4 Study to Evaluate Efficacy, Safety and Mucosal Healing of Early Versus Late Use of Vedolizumab in Ulcerative Colitis: the LOVE-UC Study (LOw Countries VEdolizumab in UC Study)
Brief Title: An Open Label Phase 4 Study to Evaluate Efficacy of Early Versus Late Use of Vedolizumab in Ulcerative Colitis
Acronym: LOVE-UC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Geert D'Haens (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor-Investigator, Geert D'Haens, Coordinating Sponsor Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-100756
Record Dates: First submitted 2015-08-27; First posted 2016-01-06 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early UC (Other): Patients with 'early UC' defined as disease duration < 4 years and no other treatments than aminosalicylates and/or corticosteroids
  Interventions: Drug: Vedolizumab 300 mg
- Late UC (Other): Patients with 'late UC' defined as active disease despite treatment with immunosuppressives (IS) and/or anti-TNF. Patients wih intolerance to IS AND anti-TNF will also be allowed in the latter group.
  Interventions: Drug: Vedolizumab 300 mg

INTERVENTIONS:
Drug: Vedolizumab 300 mg — Open-label VEDOLIZUMAB 300 mg at week 0,2,6, 14, 22, 30, 38, 46
  Other Names: Entyvio

SUMMARY:
This multi-centre open label study will involve a minimum of 120 patients in 2 cohorts: 60 patients with 'early UC' defined as disease duration < 4 years and no other treatments than aminosalicylates and/or corticosteroids and 60 patients with 'late UC' defined as active disease despite treatment with immunosuppressives (IS) and/or anti-TNF. Patients wih intolerance to IS AND anti-TNF will also be allowed in the latter group. Participants will be treated with 12 months of open label vedolizumab and undergo monitoring of endoscopic, histological and clinical disease parameters. No randomization or blinding will be performed but the study management will make sure recruitment in either study group is comparable for number and profile of patients (extent of disease and on/off corticosteroids).

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic inflammatory disease of the colon. Symptoms include bloody diarrhea, weight loss, and fever. There is no known cause or cure for UC. The aim of current UC treatments is to induce and maintain remission, to reduce the need of corticosteroids and avoid colectomy.

Treatment options include 5-Aminosalicylates (5-ASA), systemic and/or topical corticosteroids, purine analogues (6-mercaptopurine and azathioprine), anti-TNF antibodies and surgery. In 2013, results from the GEMINI I, phase 3, randomized controlled trial demonstrated the efficacy of vedolizumab (VDZ) in inducing and maintaining remission in adult patients with active UC.

VDZ (MLN0002 or MLN02), inhibits the interaction between α4β7 integrin on memory T and B cells and mucosal addressin cell adhesion molecule-1 expressed on the vascular endothelium of the gut and has been shown to be effective in both inducing and maintaining clinical remission in UC.

With other (anti-TNF) biologics, outcomes have usually been better if the treatment was started earlier in the disease course and if the patients had not been exposed to prior antibody treatments. Therefore, it appears appropriate and desirable to test the potency of vedolizumab in an earlier phase of UC. Indeed, also with vedolizumab patients previously exposed to biologics appear to have lower success rates with vedolizumab, so a position earlier in the disease course would most likely lead to better outcomes.

This is an investigator-initiated open label study of VDZ therapy in 2 distinct populations of UC patients with active disease: 1. patients who have been diagnosed < 4 years ago and who only have been exposed to aminosalicylates and corticosteroids and 2. patients who have been exposed to immunomodulators and/or anti-TNF agents in addition to steroids and aminosalicylates.

VDZ has been shown to be efficacious at inducing and maintaining remission in UC. However, data about the endoscopic and histological effects of VDZ in 'early UC' are lacking. Therefore, the investigators propose to perform an interventional study in early and late UC patients including endoscopic and histological assessment

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the subject is capable of understanding and complying with protocol requirements.
2. The subject signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Age 18 to 80
4. Male or non-pregnant, non-lactating females. Females of child bearing potential must have a negative serum pregnancy test prior to randomization, and must use a hormonal (oral, implantable or injectable) or barrier method of birth control throughout the study. Females unable to bear children must have documentation of such in the source records (i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since the last menstrual period]).
5. Established diagnosis of ulcerative colitis with histopathological confirmation available in the record of the patient.
6. Moderate to severe active UC (total Mayo score > 6) with objective evidence of inflammation that can be visualized on endoscopy. All endoscopies will be video-taped for later review, rereading and quality assurance. Patients must have an endoscopic Mayo score of 2 or 3.
7. Anti-TNF discontinued for at least 6 weeks
8. Written informed consent must be obtained and documented

GROUP 1 (EARLY UC)

1. Diagnosis of UC < 4 years prior to enrollment confirmed by clinical, endoscopic and histopathological evidence.
2. Demonstrated failure to respond to aminosalicylates or intolerance to aminosalicylates and: failure to respond to topical or systemic corticosteroids or intolerance to corticosteroids or: need for > 1 course of steroids per year or: steroid dependency at any dose and additionally, but not mandatory, lack of efficacy of thiopurines or intolerance to thiopurines (azathioprine, 6-mercaptopurine or 6-thioguanine) (any duration). Patients who are using thiopurines at screening must have used them for > 3 months (last 4 weeks at stable dose).

GROUP 2 (LATE UC)

1. Diagnosis of UC confirmed by clinical, endoscopic and histopathological evidence.
2. Demonstrated failure to respond to aminosalicylates or intolerance to aminosalicylates and: failure to respond to at least 3 months of thiopurines (TP) or intolerance to TP and: failure to respond to at least 1 anti-TNF or intolerance to anti-TNF or loss of response to at least 1 anti-TNF. Loss of response to anti-TNF is defined as recurrence of symptoms during maintenance dosing following prior clinical benefit.

May continue stable dose of conventional therapies for Inflammatory Bowel Disease ( IBD) including aminosalicylates and thiopurines and corticosteroids. Steroids will be tapered by protocol by week 14. Anti-TNF must be discontinued for > 6 weeks.

Exclusion Criteria:

1. Prior treatment with vedolizumab.
2. Contraindication for endoscopy.
3. History of colonic dysplasia/cancer
4. Extensive colonic resection, i.e. subtotal or total colectomy with <15 cm colon remaining
5. Received other biologics within the last 4 weeks of baseline
6. Use of 5-ASA or corticosteroid enemas/suppositories within 2 weeks of enrollment
7. Chronic hepatitis B or C infection
8. Evidence of or treatment for C. difficile infection or other intestinal pathogen at screening within 4 weeks prior to enrollment
9. Active or latent tuberculosis
10. Conditions which in the opinion of the investigator may interfere with the subject's ability to comply with the study procedures.
11. Received any investigational drug in the past 30 days or 5 half-lives, whichever is longer.
12. Positive progressive multifocal leukoencephalopathy (PML) subjective symptom checklist before enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-07; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Clinical and endoscopic remission | Change in Mayo score from baseline to week 26
  Defined as a Mayo Clinic score ≤2 and no subscore >1

SECONDARY OUTCOMES:
Proportion of patients with endoscopic response | Week 26 and week 52
  Change in endoscopic Mayo score of 1 or more than 1
Proportion of patients with clinical response | 52 weeks
  Mayo score < 6
Proportion of patients with clinical remission | 52 weeks
  Mayo Clinic score ≤2 and no subscore >1
Proportion of patients with corticosteroid- free clinical remission | 52 weeks
  Mayo remission score ≤2 and no subscore >1
Proportion of patients with normalized serum C-reactive protein (CRP) | 52 weeks
  Normal CRP
Proportion of patients with 25%, 50% and 75% reduction in the Geboes histology score | At week 26 and week 52
  Geboes score reduction
Proportion of patients with sustained clinical response | After week 10.
  A Mayo score < 6
Proportion of patients with sustained clinical remission | After week 10.
  Mayo Clinic score ≤2 and no subscore >1.
Proportion of patients that need to be hospitalized | 52 weeks
  hospitalization
Quality of life measured by Inflammatory Bowel Disease Questionnaire ( IBDQ ) | At enrollment, week 26 and week 52
  Questionnaire
Work productivity Index | At enrollment, week 26 and week 52
  Questionnaire
Serum concentrations of vedolizumab and antibodies to vedolizumab | Before every infusion
  through concentration
Quality of life measured by and Euroquol | At enrollment, week 26 and week 52
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Geert D'Haens, Prof., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (20):
- Belgium (12):
  - Imeldahospital, Bonheiden
  - ULB Erasme, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - AZ Sint-Lucas, Ghent
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - Leuven AcademicHospital, Leuven
  - CHC Clinique Saint-Joseph, Liège
  - CHU Liege, Liège
  - ZNA Jan Palfijn, Merksem
  - AZ Damiaan, Ostend
  - AZ Delta- Roeselare, Roeselare
- Hungary (3):
  - Semmelweis University, Budapest
  - University of Debrechen, Debrecen
  - University of Szeged, Szeged
- Netherlands (5):
  - Academic Medical Center, Amsterdam
  - OLVG, Amsterdam
  - Ziekenhuis Gelderse Vallei, Ede
  - Radboud UMC, Nijmegen
  - Erasmus MC, Rotterdam